CLINICAL TRIAL: NCT04518904
Title: Establishment of a Prognosis Prediction Model and Scoring Criteria of Pulmonary Contusion Caused by Severe Thoracic Trauma
Status: Completed | Type: Observational
Sponsor: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Responsible Party: Principal Investigator, Lei Wang, attending doctor of Thoracic surgery, Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Other Study IDs: ynhg201919
Record Dates: First submitted 2020-08-17; First posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Pulmonary Contusion , Chest Trauma , Prediction Model
Keywords: pulmonary contusion; severe chest trauma; prediction model
MeSH Terms: conditions — Thoracic Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group of poor prognosis: In this group,the patients had suffered from systemic infection,pulmonary complications or died.
- Group of good prognosis: In this group,the patients were safely discharged without complications.

INTERVENTIONS:
Other:

SUMMARY:
Pulmonary contusion caused by severe thoracic trauma is a complex disease. Some patients may be secondary to severe complications such as pulmonary infection or even acute respiratory distress syndrome. At present, there have been no reports on related studies based on Chinese population. In this study, 800 patients with pulmonary contusion will be retrospectively investigated to determine the risk factors and independent risk factors of their poor prognosis, and to construct a prognosis prediction model and scoring criteria.

ELIGIBILITY:
Inclusion Criteria:

Chinese patients aged 18 to 80 years,severe chest trauma (flail chest, more than 4 rib fractures without flail chest, multiple anterior rib fractures with sternal fractures, bilateral fractures, severely displaced sternal fractures),pulmonary contusion.

Exclusion Criteria:

Patients were excluded if they had a history of tuberculosis, heart failure,respiratory failure,severe brain injury(GSC score < 15),loss of consciousness, spinal fracture complicated with paraplegia,abdominal trauma requiring surgical intervention,shock.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 800 cases of patients were hospitalized from 2014 to 2019.All patients were Chinese.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
To build a prognostic prediction model and standard scoring system for pulmonary contusion caused by severe chest trauma | 2020.1-2020.6,enter data by protocol, statistical analysis,
  In this study, 800 patients with pulmonary contusion will be retrospectively investigated to determine the risk factors and independent risk factors of their poor prognosis, and to construct a prognosis prediction model and scoring criteria.

IPD SHARING:
Plan to Share IPD: No